CLINICAL TRIAL: NCT00588939
Title: Confocal Laser Microscopy in Non Erosive Reflux Disease
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenneth K. Wang, VanCleve Professor of Gastroenterology Research, Mayo Clinic
Other Study IDs: 07-006186
Record Dates: First submitted 2007-12-22; First posted 2008-01-09 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Acid Reflux Disease; Heartburn
Keywords: reflux; heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — esophageal biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I: participants with symptoms of acid reflux disease (heartburn)
  Interventions: Device: Cell~vizio (Laser connfocal microscopy)

INTERVENTIONS:
Device: Cell~vizio (Laser connfocal microscopy) — completed during endoscopy
  Other Names: Mauna Kea Cellvizeo

SUMMARY:
Heartburn or reflux disease affects about 20% of Americans. 50 - 70% of people who have endoscopy for reflux disease have a normal appearing esophagus. Confocal Laser Microscopy allows us to see changes in the cells not visable during routine endoscopy. Whe goal of this study is to identify the use of this new technique in diagnosing reflux in patients who have normal appearing esophagus.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) remains a major problem in the United States affecting about 20% of Americans. Upper endoscopy (EGD) is commonly used to diagnose and grade GERD based on mucosal breaks and erosions. It is now evident from multiple studies however that the majority of GERD patients (50-70%) have negative EGDs.These patients are refered to as "Non Erosive Reflux Disease" (NERD) patients.Confocal Laser Microscopy (CLM) is a new endoscopic technique that offers the advantage of detecting histologic changes during real time endoscopy and thus can diagnose NERD. We thus propose to study the sensitivity and specificity of CLM in predicting NERD. We hypothesize that CLM can reliably diagnose NERD in the appropriate clinical setting based on intrapapillary capillary loop patterns. This will be a pilot study after which a randomized trial will evaluate the reversibility of these changes after PPI therapy as seen by CLM

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years to 85 years old who are referred for an upper endoscopy for symptoms of reflux disease
2. Patients who are able to give informed consent

Exclusion Criteria:

1. Patients with a history of Erosive esophagitis
2. Patients with a history of Barrett's esophagus
3. Patients who on upper endoscopy have any current evidence of erosive esophagitis, Barrett's esophagus or varices
4. Patients who are unable or unwilling to undergo endoscopic evaluation
5. Patients who are unable to give informed consent
6. Patients with a known coagulopathy who are unable to be off therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age 18 - 65 years symptoms of acid reflux disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess the sensitivity, specificity, negative and positive predictive value of CLM in diagnosing NERD | at time of procedure

SECONDARY OUTCOMES:
To assess the additional charges of implementing CLM in EGD | at time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Wang, MD, Study Director — Mayo Clinic; Rami Badreddine, MD, Principal Investigator — Malyo Clinic Rochester
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States